CLINICAL TRIAL: NCT02441075
Title: 70% Ethanol for Decontamination of CVL Exposed to Calcineurine Inhibitors Version 1.0, 1/9/2014
Acronym: 70% EtOH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Daisy Foundation (Other)
Responsible Party: Principal Investigator, Rajinder Bajwa, Principal Investigator, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-00028
Record Dates: First submitted 2015-04-30; First posted 2015-05-12 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Hematopoietic Stem Cell Transplant; GVHD
Keywords: patients; BMT; cyclosporine; tacrolimus; HSCT
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 70% Ethanol (Experimental): The study will use 70% ethanol lock in the CVLs. A 2ml 70% ethanol lock will be instilled into the white lumen of the CVL for 2 hours. At the end of 2 hours, the ethanol will be withdrawn; the CVL lumen flushed with normal saline, and the CVL would be available for normal use for that day.
  Interventions: Other: 70% Ethanol

INTERVENTIONS:
Other: 70% Ethanol — the study will use 70% ethanol lock in the CVLs. A 2ml 70% ethanol lock will be instilled into the white lumen of the CVL for 2 hours. At the end of 2 hours, the ethanol will be withdrawn; the CVL lumen flushed with normal saline, and the CVL would be available for normal use for that day.

SUMMARY:
This is for a study for patients that will be undergoing hematopoietic stem cell transplant (HSCT). For HSCT, patients will need a double lumen central venous line (CVL). One of the most common complications after an HSCT is Graft Versus Host Disease (GVHD).Tacrolimus or Cyclosporine along with methotrexate are used together in order to prevent GVHD. Normally these medications are given via the white lumen and blood is drawn via the unexposed red lumen to check the blood level of these medications. If these drugs are accidentally given via the wrong lumen (line) it could cause blood levels to be falsely high. This error could lead to the patient having to have peripheral blood draws that cause pain. The investigators are proposing adding an ethanol lock to your lumens (lines) to see if this would help clean the lines therefore preventing errors in blood tests and blood draws. An ethanol lock is a 70% alcohol which is injected into the CVL lumen and stays within the CVL as the CVL is capped.

DETAILED DESCRIPTION:
As cyclosporine and tacrolimus are both oil based medications and ethanol (70% alcohol) can dissolve oil, the investigators hypothesize that an alcohol lock instilled into the lumen of the CVL will be able to dissolve and leach out the oil based CNI adhering to the inside lumen of the CVL catheter, thus decontaminating it. The safety of using ethanol via CVL is already proven over the last many years. A study performed with neonates resulted in no adverse effects when using ethanol locks, proving that their use is safe for the pediatric population. Ethanol has been used as locks for disinfecting CVLs infected with a broad range of microorganisms in pediatrics. It has also been useful in treating catheter occlusions caused by Lipid formation. By placing a 70% ethanol lock for two hours in the contaminated lumen, it has shown to degrade the biofilm and fat formation allowing for further use of the CVL used 70 % ethanol locks and did not find any reductions in mechanical integrity of polyetherurethane or silicone catheters exposed for as long as 10 weeks. Also, no structural integrity complications have been found in the literature along with no evidence of systemic toxicity with the use of ethanol locks. A retrospective study on PICU patients who had received ethanol locks for 12-24 hours per lumen and a repeat lock when venous access was not limited, flushed 0.2-1mls of ethanol through the catheter at the end of the dwell instead of withdrawing the lock. Sixteen patients who received five daily ethanol lock treatments in succession, had liver enzymes measured and only two patients had mildly elevated transaminases, but these levels were not significant from their baseline levels. There were also no reports from the nurses of any patient complaints or side effects. The study stated that when larger volumes in which they classified as 2.3mls of ethanol are flushed through the central line, patients have reported flushing, light-headedness, headache, nausea and dyspnea. Only 2mls of ethanol will be administered in this study, and the ethanol lock will be withdrawn prior to drawing the levels. Therefore, no side effects are expected.

ELIGIBILITY:
Inclusion Criteria:

* All patients' ages 3 months to 30 years will be eligible for the study.
* All patients undergoing an allogeneic HSCT and receiving intravenous cyclosporine or tacrolimus through a CVL will be eligible.

Exclusion Criteria:

* Patients who are hemodynamically compromised or needing intensive care in the ICU.
* Family/patient not willing to sign an informed consent.

Ages: 3 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: Serum Levels | 18 months
  Serum levels from both lumens will be compared after 2-hour ethanol lock placements. If the mean serum levels drawn at 8pm from both lumens are equivalent, the intervention will be considered effective.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States